CLINICAL TRIAL: NCT04444791
Title: Chinese Pregnant Woman Cohort Study (Offspring Follow-up)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Yu Jiang, School of Public Health, Peking Union Medical College
Other Study IDs: PUMCPublicHealth
Record Dates: First submitted 2020-06-20; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy Related; Pregnancy Disease; Pregnancy; Infant Development; Risk Factor; Infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: This cohort study only set up one group. The habits and health status of mothers and their offspring will be followed up and observed. The participants will be divided into more than one group according to the variables (e.g. age, physical activity, dietary patterns, sleep quality.).

SUMMARY:
Purpose: To investigate the growth and development status for children of 1 ~ 3 years old in China, and to explore and analyze the influencing factors of infant growth. Mother's health status would also be investigated simultaneously.

Methods and analysis: This is a multicenter prospective cohort study. Participants were all from the Chinese Pregnant Women Cohort Study (CPWCS), which is a multicenter prospective cohort study we conducted before. In simple terms, pregnant women during the first trimester (5~13 weeks' gestational age) were included from 25 July 2017 to 26 November 2018. Related information were collected by electronic self-administered questionnaire, including general information, environmental exposure assessment, physical activity assessment, dietary and nutritional assessment, depression assessment, sleep quality assessment and economic burden assessment. Subsequently, objective medical information, obstetric and neonatal outcomes were collected through hospital information system (HIS).

To further assess the mothers' and infants' health status, a new multicenter prospective cohort study, including more than 1000 participants of the CPWCS from 5 hospitals of 5 different provinces in China, will be conducted. Through the electronic self-administered questionnaire surveys and laboratory testing methods, information about infants' feeding, sleeping, defecating, oral health, early development and common allergic diseases will be collected. And we will also assess mothers' current health habits and status, such as sleeping, diet, anxiety, physical activity, and oral health. SAS statistical software will be used for data analysis.

Ethics and Dissemination Permission for the study was obtained from Chinese Academy of Medical Sciences and Peking Union Medical College. Ethics approval was obtained from the Ethics Review Committee of Department of Scientific Research, School of Basic Medicine, Peking Union Medical College, Beijing, China. The results will be published in peer-reviewed journals or disseminated through conference presentations.

ELIGIBILITY:
Inclusion Criteria:

1. participated in the CPWCS and were pregnant women included in the previous cohort;
2. the baseline, first trimester, delivery outcomes, and neonatal outcomes data in the CPWCS were complete;
3. live birth and singleton in the CPWCS;
4. participate in the CPWCS-OF with child born in the CPWCS willingly;
5. able to complete the questionnaire;
6. resident in the study area;
7. signed the informed consent.

Exclusion Criteria:

1. subjects not included in the CPWCS;
2. incomplete data in either of baseline, first trimester, delivery outcomes, and neonatal outcomes in the CPWCS;
3. pregnancy outcomes in the CPWCS were not singleton (abortion, stillbirth, twins, multiple births);
4. no longer resident in the study area;
5. the child has died;
6. the mother currently has mental problems and cannot cooperate well with the research.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In the Chinese Pregnant Women Cohort Study (CPWCS), more than 9000 pregnant women were recruited from 25 July 2017 to 26 November 2018 during their routine antenatal check at the first trimester. Five hospitals of 5 different provinces in China with certain working foundation, good cooperation and high follow-up rate of pregnant women in the CPWCS were selected as study sites for the new cohort of the Chinese Pregnant Women Cohort Study-Offspring Follow-up (CPWCS-OF). From these 5 hospitals, mothers with the baseline information, first trimester questionnaire, delivery outcomes, and neonatal outcomes data completed, and had live birth and singleton were included. According to the inclusion and exclusion criteria, 1978 mothers with their infants were selected as the research objects.
Sampling Method: Probability Sample
Enrollment: 1978 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Infants' and young children's feeding situation | 2020.8.1-2020.12.1
  The mother will report these questions.
Infants' sleeping conditions | 2020.8.1-2020.12.1
Infants' defecation situation | 2020.8.1-2020.12.1
Infants' oral development | 2020.8.1-2020.12.1
Infants' early development | 2020.8.1-2020.12.1
Mother' knowledge of infant oral health care | 2020.8.1-2020.12.1
Infants' physical health (asthma, allergies, autism) | 2020.8.1-2020.12.1

SECONDARY OUTCOMES:
Mothers' physical activity | 2020.8.1-2020.12.1
Mothers' dietary patterns | 2020.8.1-2020.12.1
Mothers' lifestyle (smoking, sleeping) | 2020.8.1-2020.12.1
Mothers' anxiety condition | 2020.8.1-2020.12.1
Mothers' oral health | 2020.8.1-2020.12.1

CONTACTS AND LOCATIONS:
Locations (1):
- School of Public Health, Peking Union Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lyu T, Chen Y, Zhan Y, Shi Y, Yue H, Liu X, Meng Y, Jing A, Qu Y, Ma H, Huang P, Man D, Li X, Wu H, Zhao J, Shan G, Jiang Y. Cohort profile: the Chinese Pregnant Women Cohort Study and Offspring Follow-up (CPWCSaOF). BMJ Open. 2021 Mar 23;11(3):e044933. doi: 10.1136/bmjopen-2020-044933. PMID 33757952